CLINICAL TRIAL: NCT05948150
Title: The Effect Of Breastfeedıng Pıllow On Breastfeedıng Self- Effıcacy And Postnatal Comfort In Prımıparous Postpartum Women Who Gave Bırth By Caesarean Sectıon
Brief Title: The Effect of Breastfeeding Pillow on Breastfeeding Self-Efficacy and Postpartum Comfort in Women Who Had Cesarean
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ataturk University (Other)
Responsible Party: Principal Investigator, İltifat Hümeyra DİNÇ, Research Assistant, Ataturk University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: AtaturkU
Record Dates: First submitted 2023-06-24; First posted 2023-07-17 (Actual); Last update posted 2023-07-17 (Actual); Status verified 2023-07

CONDITIONS: Cesarean Section; Dehiscence; First Birth
Keywords: Breastfeeding; Exclusive Breast Milk; Patient Comfort; Self-efficacy
MeSH Terms: conditions — Breast Feeding

STUDY DESIGN:
Intervention Model Description: Quantitative
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group not to use a breastfeeding pillow (Experimental): In this arm, individuals are not provided with a breastfeeding pillow.
  Interventions: Other: not using a breastfeeding pillow
- breastfeeding pillow group (Experimental): In this arm, breastfeeding pillows are used for individuals
  Interventions: Other: using a breastfeeding pillow

INTERVENTIONS:
Other: using a breastfeeding pillow — To make the breastfeeding pillow group use the breastfeeding pillow from the 8th hour in the postnatal period and to make evaluations at 24 and 48 hours
  Arms: breastfeeding pillow group
Other: not using a breastfeeding pillow — The non-breastfeeding pillow group was evaluated at 24 and 48 hours without the use of a breastfeeding pillow
  Arms: group not to use a breastfeeding pillow

SUMMARY:
The research is a randomised controlled experimental study. It was conducted to examine the effect of breastfeeding pillow on breastfeeding self-efficacy and postnatal comfort in primiparous puerperas who gave birth by caesarean section. The answers to the questions "Is the breastfeeding pillow effective on breastfeeding self-efficacy in primiparous puerperium giving birth by caesarean section?" and "Is the breastfeeding pillow effective on comfort during breastfeeding in primiparous puerperium giving birth by caesarean section?" are investigated. The puerperas in the experimental group were allowed to use a breastfeeding pillow during breastfeeding and evaluated at 24th and 48th hours. Puerperas in the control group continued routine breastfeeding and did not use a breastfeeding pillow. They were evaluated at 24th and 48th hours.

ELIGIBILITY:
Inclusion Criteria:

* Graduated from primary school
* No communication problems
* The desire to breastfeed your baby,
* The mother and the baby do not have any health condition that may prevent breastfeeding,
* First pregnancy,
* Having given birth at 37> 37 weeks of gestation,
* Having a baby weighing at least 2500 g,
* Over 18 years of age,
* Caesarean section with a single healthy baby

Exclusion Criteria:

* having given birth more than once
* Under 18 years of age
* communication problems
* unhealthy baby birth

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2022-11-29 (Actual); Primary Completion 2023-05-30 (Actual); Study Completion 2023-06-23 (Actual)

PRIMARY OUTCOMES:
Increasing breastfeeding self-efficacy by using a nursing pillow | 48 hours
  Increasing breastfeeding self-efficacy in puerperant women who gave birth by using a nursing pillow
Increasing postpartum comfort by using a nursing pillow | 48 hours
  Increasing postpartum comfort in postpartum women who gave birth by using a nursing pillow

CONTACTS AND LOCATIONS:
Overall Officials: İltifat H Dinç, Principal Investigator — humeyra.dinc@erzincan.edu.tr
Locations (1):
- Erzincan Binali Yıldırım University Mengücek Gazi Training and Research Hospital, Erzincan, Turkey (Türkiye)